CLINICAL TRIAL: NCT04198467
Title: Randomized Controlled Study to Compare Safety and Efficacy of Intra Articular Administration of Platelet Rich Plasma Versus Hyaluronic Acid as Placebo in Patients With Osteoarthritis of Knee
Brief Title: To Evaluate the Optimum Dose of Platelet Rich Plasma in Knee Osteoarthritis and Compare Efficacy With Hyaluronic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Himanshu Bansal Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HimanshuBansalF
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; hylan

STUDY DESIGN:
Intervention Model Description: 182 patients screened, 100 were considered eligible for the study and were randomized. The most common reason for exclusion was either the lack of radio graphic evidence of knee OA or the presence of severe disease with JSW less than 2 mm at the narrowest point.
  Out of the 100 randomized patients, roughly equal numbers, six patients in PRP and 7 in placebo, did not complete the study. Reasons for withdrawal were personal,inefficacy, or adverse event as an increase in pain.
Who Masked: Participant, Investigator
Masking Description: Hyaluronic acid as placebo both patient and investigator blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP (100billion platelets) (Experimental): platelet rich plasma having 100 billion platelets in 10 ml plasma prepared from 60 ml blood
  Interventions: Biological: Platelet rich plasma
- hyaluronic acid (Placebo Comparator): Four ml of high-molecular-weight hyaluronic acid (HMWHA) with a concentration of 22mg/ml
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: Platelet rich plasma — Platelet rich plasma : 100 billion platelets in 10 ml of plasma(PRP) administered intra-articular
  Other Names: PRP
  Arms: PRP (100billion platelets)
Drug: Hyaluronic Acid — Hyaluronic acid :Four ml of high-molecular-weight hyaluronic acid with a concentration of 22mg/ml injected intra-articular
  Other Names: SYNVISC
  Arms: hyaluronic acid

SUMMARY:
Randomized, Double-blind, 12-month, placebo-controlled study was conducted on 100 outpatients . Intervention platelet rich plasma( PRP) prepared from 60 ml of blood by adding novel step of filtration to manual centrifuge step to achieve 7 times concentration. the efficacy was compared with administration of hyaluronic acid. Subjective Womac scores ,6 min pain free walking distance as well objective assessments MRI ,synovial fluid assessments were made out .Absolute counts of platelets as dose was evaluated to be effective in alleviating symptoms in early knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) causes substantial physical disability that limits a person ability to indulge in daily activities. OA related disability has been affecting millions of older adults throughout the world, and the number has almost doubled in 2019.

Though the process of OA could not be reversed, efficient management strategies could help in minimizing primary pain with physical exercises, surgical procedures, and medications.

Prolonged use of nonsteroidal anti-inflammatory drugs (NSAIDs) has been dramatically associated with mild to severe side effects, limiting its continuous use. Chondro-protective agents (CPAs) have been proven to provide only minimal symptomatic benefit. Platelet-rich plasma (PRP) has emerged as a supreme therapy in OA knee however exact dose ,preparation and duration of benefit still remains unclear.

Study was undertaken to demonstrate the potential of leukocyte depleted PRP in cartilage repair of knee OA using WOMAC scores as subjective assessment tool.

Our research also evaluated objective criteria ing joint space width (JSW),cartilage thickness on MRI, Ultrasound that would improve knee joint function in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who fulfilled the clinical and radiological criteria set by the American College of Rheumatology for the diagnosis of symptomatic primary knee OA, with pain Visual Analogue Scale (VAS) score of >3 in the previous month. In cases where both the knees were symptomatic, the knee which was comparatively more painful was considered.

Exclusion Criteria:

1. Evidence of secondary knee OA because of injury, inflammatory or metabolic rheumatic disease, or osteonecrosis;
2. Prior intra-articular injection of hyaluronic acid (HA), including lavage and corticosteroids within the previous three months;
3. Severe knee OA, with JSW <1 mm, or surgery required on the evaluated knee in the year
4. Patients with clinically significant systemic disease.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
changes in womac score | baseline,1 month,3 months,6 months, and 1year
  WOMAC, a widely used measure to assess patients' pain, joint mobility, and physical disability evaluates three dimensions, pain, stiffness, and physical function, with 5, 2, and 17 questions, respectively. The total maximum score is 96 and minimum, 0
changes in cartilage thickness as assessed on 1.5 T MRI | baseline and at one year
  Using the 1.5-T field strength with standard MRI acquisition protocols, MRI was performed of each joint individually in coronal, sagittal, and transverse planes. The maximum thickness of the cartilage at posterior,meniscal and patellar level measured at the midsagittal plane through the medial condyle was considered. The medial femoral cartilage of the affected knee was chosen for measurement.

SECONDARY OUTCOMES:
changes in joint space width | baseline and at 12months
  Patients were radiographed in a weight-bearing position, joints fully extended, standing at 1 m from the X-ray source20. The width was measured at the narrowest point of the Joint (JSW)
changes in cartilage thickness as assessed by ultrasonically. | baseline ,6 months and at 12 months
  Having the patients sit with flexed knees,The articular cartilage of the medial femoral condyle was evaluated with a starting point at the level of intercondylar notch to the medial border of the medial condyle by an ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: himanshu bansal, ms, Principal Investigator — anupam hospital rudrapur uttrakhand

IPD SHARING:
Plan to Share IPD: Yes
Anyone interested, Researcher ,Patient or Institute can contact and we would gladly assist him with all information. Nothing is hidden
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be always available to anyone interested
Access Criteria: Anyone interested, Researcher ,Patient or Institute can access data anytime.
URL: http://www.drhbf.org

REFERENCES:
- [Result] Riboh JC, Saltzman BM, Yanke AB, Fortier L, Cole BJ. Effect of Leukocyte Concentration on the Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis. Am J Sports Med. 2016 Mar;44(3):792-800. doi: 10.1177/0363546515580787. Epub 2015 Apr 29. PMID 25925602
- [Result] Paterson KL, Nicholls M, Bennell KL, Bates D. Intra-articular injection of photo-activated platelet-rich plasma in patients with knee osteoarthritis: a double-blind, randomized controlled pilot study. BMC Musculoskelet Disord. 2016 Feb 9;17:67. doi: 10.1186/s12891-016-0920-3. PMID 26861957
- [Result] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403